CLINICAL TRIAL: NCT02618590
Title: Which Treatment Strategy is Best in Non-small Cell Lung Cancer Patients Harboring EGFR Mutant Type After First/Second Line EGFR-TKI Failure, a Retrospective Study
Brief Title: A Retrospective Study About Treatment Strategy After First/Second Line EGFR-TKI Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, Associate Professor/Associate chief physician, Sun Yat-sen University
Other Study IDs: 2015-FXY-029-内科
Record Dates: First submitted 2015-08-22; First posted 2015-12-01 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: non-small cell lung cancer; EGFR mutant type; first/second line EGFR-TKI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a multi-center retrospective study, designing to access the best treatment strategy in non-small cell lung cancer (NSCLC) patients harboring EGFR mutant type after first/second line EGFR-TKI failure. The study end point is Progression Free Survival 2 (PFS2), which is defined as the time period from Progression Disease 1(PD1) to Progression Disease 2(PD2). PD1 is defined as the first tumor progression time from taking EGFR-TKI evaluated by Recist 1.1 criterion, and PD2 as the second tumor progression time after EGFR-TKI failure no matter what second/third line treatment was, PD2 is also evaluated by Recist 1.1 criterion.

ELIGIBILITY:
Inclusion Criteria:

* Patients who was confirmed stage IV (according to International Association for the Study of Lung Cancer（IASLC） TNM staging, 2009) non-small cell lung cancer (NSCLC) by histology or cytology between year 2009 to 2013, harboring EGFR mutant type (19 and/or 21 exon mutation).
* Appraisable disease, that is there must be at least one lesion with the longest diameter>10mm according to Recist 1.1 criterion (by contrast CT).
* Patients who take EGFR-TKI as first/second line therapy.

Exclusion Criteria:

* Patients who has taken EGFR-TKI before.
* Patients who take EGFR-TKI as third or more line.
* Patients who take EGFR-TKI concurrent with chemotherapy or other anti-tumor drug.
* The evaluated lesions has treated with radiotherapy before or concurrent with EGFR-TKI.
* Patients whose EGFR expression is positive by immunochemical and/or EGFR amplification is positive by Fluorescence In Situ Hybridization(FISH), without mutation detection evidence.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with stage IV non-small cell lung cancer (NSCLC) harboring EGFR mutant type (19 and/or 21 exon mutation), and took EGFR-TKI as first/second line therapy.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival 2 (PFS2) | 6 months

SECONDARY OUTCOMES:
overall survival (OS) | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: li-kun Chen, doctor, Principal Investigator — associate chief physician
Locations (1):
- Sun Yat-sen University of cancer center, Guangzhou, Guangdong, China